CLINICAL TRIAL: NCT02821819
Title: Random-start Ovarian Stimulation in Egg-donors (ROSE) Trial: a Self-controlled Study
Brief Title: Random-start Ovarian Stimulation in Egg-donors (ROSE)
Acronym: ROSE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficult recruitment
Sponsor: Instituto Bernabeu (Other)
Responsible Party: Principal Investigator, Juan Carlos Castillo, Md. PHd., Instituto Bernabeu
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IB012016
Record Dates: First submitted 2016-06-19; First posted 2016-07-04 (Estimated); Results first posted 2019-08-19 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-07

CONDITIONS: Infertility
Keywords: ovarian stimulation; random; egg donation; antagonist; gnrh agonist trigger
MeSH Terms: conditions — Infertility | interventions — Ovulation Induction; Gonadotropins; LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Random start ovarian stimulation (Experimental): Egg-donors will be assigned to random start ovarian stimulation: During follicular phase starting at day 5,7,9,11 or 13 of the menstrual cycle and during luteal phase at luteinizing hormone (LH) peak +3,+5,+7,+9 or +11. They will receive urinary follicle stimulating hormone (FSH) 150-225 International units / daily (IU/d) and five days later the gonadotropin-releasing hormone (GnRH) antagonist: cetrorelix acetate 0,25 mg/d will be added until achieving criteria for receiving triptorelin 0,2 mg to induce final follicular maturation. Egg collection will take place 36 hours later.
  Interventions:
  * Random start ovarian stimulation
  * Gonadotrophins: Urinary FSH 150-225 IU/d
  * GnRH antagonists: Cetrorelix 0,25 mg/d
  * GnRH agonist for triggering: Triptorelin 0,2 mg single dose
  Interventions: Other: Random start ovarian stimulation; Drug: Gonadotrophins; Drug: GnRH antagonist; Drug: GnRH agonist

INTERVENTIONS:
Other: Random start ovarian stimulation — Egg-donors will start ovarian stimulation randomly at different moments throughout the menstrual cycle.
  Other Names: Ovarian stimulation
Drug: Gonadotrophins — Urinary FSH 150-225 IU/d
  Other Names: Ovarian stimulation
Drug: GnRH antagonist — Cetrorelix acetate 0,25 mg/d starting five days after ovarian stimulation
  Other Names: Ovarian stimulation
Drug: GnRH agonist — GnRH agonist triggering with triptorelin 0,2 mg for final follicular maturation.
  Other Names: Final follicular maturation

SUMMARY:
The purpose of this prospective single-center study is to evaluate the laboratory outcome after random start ovarian stimulation in oocyte donors. The study will be performed in egg-donors but this type of treatment has the potential to be implemented in general infertility population.

DETAILED DESCRIPTION:
The study group will start ovarian stimulation randomly in different moments throughout the menstrual cycle.

Randomization will take place on day 2-3 of the menstrual cycle, according to a list of random allocation of treatments and egg-donors will be assigned to random start ovarian stimulation: During follicular phase starting at day 5,7,9,11 or 13 of the menstrual cycle and during luteal phase starting at luteinizing hormone (LH) peak +3,+5,+7,+9 or +11.

Egg-donors will receive urinary follicle stimulating hormone (FSH) 150-225 IU/d in gonadotropin-releasing hormone (GnRH) antagonist protocol with cetrorelix acetate 0,25 mg/d starting five days after ovarian stimulation and a GnRH agonist trigger with triptorelin 0,2 mg to induce the final follicular maturation. Transvaginal ultrasound and serum analysis (estradiol, progesterone, LH and FSH) will be included for cycle monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women
* 18-35 years old
* FSH levels < 10 IU/liter
* Antral follicle count (AFC) > 10
* Regular cycles
* Body Mass Index (BMI) < 28
* Signed informed consent

Exclusion Criteria:

* Polycystic ovary syndrome (PCOS) patients
* Allergy to gonadotrophins
* Concomitant participation in other trial

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2018-01-12 (Actual); Study Completion 2018-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan C Castillo, Md. PhD., Principal Investigator — Instituto Bernabeu
Locations (1):
- Instituto Bernabeu, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Setting — http://www.institutobernabeu.com
- See also: Reference — http://www.ncbi.nlm.nih.gov/pubmed/27114329

RESULTS

PARTICIPANT FLOW:
Groups:
- Random Start Ovarian Stimulation: Egg-donors will be assigned to random start ovarian stimulation: During follicular phase starting at day 5,7,9,11 or 13 of the menstrual cycle and during luteal phase at luteinizing hormone (LH) peak +3,+5,+7,+9 or +11. They will receive urinary follicle stimulating hormone (FSH) 150-225 International units / daily (IU/d) and five days later the gonadotropin-releasing hormone (GnRH) antagonist will be added until achieving criteria for receiving triptorelin 0,2 mg to induce final follicular maturation. Egg collection will take place 36 hours later.
  Interventions:
  * Random start ovarian stimulation
  * Gonadotrophins: Urinary FSH 150-225 IU/d
  * GnRH antagonists: Cetrorelix 0,25 mg/d
  * GnRH agonist for triggering: Triptorelin 0,2 mg single dose
  Gonadotrophins: Urinary FSH 150-225 IU/d
  GnRH antagonist: Cetrorelix acetate 0,25 mg/d starting five days after ovarian stimulation
  GnRH agonist: GnRH agonist triggering with triptorelin 0,2 mg for final follicular maturation.
Period: Overall Study
Arm/Group | Random Start Ovarian Stimulation
Started | 15
Completed | 14
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Groups:
- Random Start Ovarian Stimulation: Egg-donors will be assigned to random start ovarian stimulation: During follicular phase starting at day 5,7,9,11 or 13 of the menstrual cycle and during luteal phase at LH peak +3,+5,+7,+9 or +11. They will receive urinary FSH 150-225 IU/d and five days later cetrorelix acetate 0,25 mg/d will be added until achieving criteria for receiving triptorelin 0,2 mg to induce final follicular maturation. Egg collection will take place 36 hours later.
  Interventions:
  * Random start ovarian stimulation
  * Gonadotrophins: Urinary FSH 150-225 IU/d
  * GnRH antagonists: Cetrorelix 0,25 mg/d
  * GnRH agonist for triggering: Triptorelin 0,2 mg single dose
  Gonadotrophins: Urinary FSH 150-225 IU/d
  GnRH antagonist: Cetrorelix acetate 0,25 mg/d starting five days after ovarian stimulation
  GnRH agonist: GnRH agonist triggering with triptorelin 0,2 mg for final follicular maturation.
Arm/Group | Random Start Ovarian Stimulation
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.2 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Mature Eggs
Description: When collected, eggs retain numerous cells (granulosa or cumulus cells) surrounding the oocyte; this structure is termed as the cumulus oocyte complex (COC). Few hours later (2-4 hs), the oocyte is denuded from these cumulus cells, allowing for a clearer observation of the maturity status (presence or absence of a metaphase II) of the oocyte. The percentage of mature eggs represents the proportion resulting from dividing the total number of COCs collected by the number of metaphase II oocytes and multiplied by 100.
Time Frame: Up to 24 hours from the oocyte collection
Measure: Mean (Standard Deviation); unit: Percentage of mature eggs
Arm/Group | Random Start Ovarian Stimulation
Number analyzed (Participants) | 15
Percentage of mature eggs | 82 (10)
Statistical Analysis 1: Comparison: Random Start Ovarian Stimulation; The sample size was calculated assuming a non-inferiority margin of 5 eggs and a standard deviation (SD) of 6.7. A unilateral alpha level of 0.05 was stablished. With the aim to show that the difference in the mean number of collected eggs will not exceed 5, a statistical power of 80% required 30 patients per group (1:1 allocation, total sample: 60); Test type: Non-Inferiority — The sample size was calculated assuming a non-inferiority margin of 5 eggs SD 6.7. A unilateral alpha level of 0.05 was stablished. With the aim to show that the difference in the mean number of collected eggs will not exceed 5, a statistical power of 80% required 30 patients per group (1:1 allocation, total sample: 60); p = 0.8, t-test, 1 sided — a priori threshold for statistical significance: <0.05; Mean Difference (Final Values) = 18, Standard Deviation 8.1; Since the number of collected eggs constitutes the main outcome of the study, the sample size was calculated assuming a non-inferiority margin of 5 eggs with an standard deviation of 6.7. A unilateral alpha level of 0.05 was stablished. With the aim to show that the difference in the mean number of collected eggs will not exceed 5, a statistical power of 80% required 30 patients per group (1:1 allocation, total sample: 60). Statistical analysis was performed using t-student test for continuous variables and chi-square test for categorical parameters. A P value of <.05 was considered significant
Statistical Analysis 2: Comparison: Random Start Ovarian Stimulation; The sample size was calculated assuming a non-inferiority margin of 5 eggs SD 6.7. A unilateral alpha level of 0.05 was stablished. With the aim to show that the difference in the mean number of collected eggs will not exceed 5, a statistical power of 80% required 30 patients per group (1:1 allocation, total sample: 60). Statistical analysis used t-student test for continuous variables and chi-square test for categorical parameters; Test type: Non-Inferiority — The sample size was calculated assuming a non-inferiority margin of 5 eggs SD 6.7. A unilateral alpha level of 0.05 was stablished. With the aim to show that the difference in the mean number of collected eggs will not exceed 5, a statistical power of 80% required 30 patients per group (1:1 allocation, total sample: 60). Statistical analysis used t-student test for continuous variables and chi-square test for categorical parameters; p = 0.8, Chi-squared — a priori threshold for statistical significance: <0.05; Mean Difference (Final Values) = 82

2. Secondary Outcome: Fertilization Rate
Description: Percentage of properly fertilized eggs after microinjection (ICSI) method
Time Frame: 24 hours after day of oocyte collection
Measure: Median (Standard Deviation); unit: Percentage of properly fertilized eggs
Arm/Group | Random Start Ovarian Stimulation
Number analyzed (Participants) | 14
Percentage of properly fertilized eggs | 71 (7.8)
Statistical Analysis 1: Comparison: Random Start Ovarian Stimulation; Test type: Non-Inferiority — Statistical analysis was performed using t-student test for continuous variables and chi-square test for categorical parameters. A P value of <.05 was considered significant; p < 0.05, Chi-squared; Median Difference (Final Values) = 71.1

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Random Start Ovarian Stimulation
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

LIMITATIONS AND CAVEATS:
Early termination. Only random-start follicular phase stimulation was completed.

01 patient was withdrawn from analysis due to protocol violation: error in administration of medication

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/19/NCT02821819/Prot_SAP_000.pdf